CLINICAL TRIAL: NCT03367468
Title: Comparison of the Different Conservative Therapy Interventions in Plantar Fasciitis
Brief Title: Conservative Therapy Interventions in Plantar Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sulenur Yildiz (Other)
Responsible Party: Sponsor-Investigator, Sulenur Yildiz, Research assistant, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06144834
Record Dates: First submitted 2017-11-10; First posted 2017-12-08 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Plantar Fascitis; Pain
Keywords: Plantar fascitis; Pain; Exercise; Physiotherapy; Quality of life
MeSH Terms: conditions — Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physiotherapy group (Active Comparator): Strengthening and stretching exercises,cross friction massage (supervised by physiotherapist) Mobilization techniques Daily usage of prescribed orthotic insole
  Interventions: Other: Exercise; Other: Mobilization
- Home exercise group (Active Comparator): Strenthening and stretching exercises Daily usage of prescribed orthotic insole
  Interventions: Other: Mobilization
- Control group (No Intervention): Follow ups Daily usage of prescribed orthotic insole

INTERVENTIONS:
Other: Exercise — Strengthening exercises ( extrinsic and intrinsic foot muscles) Stretcthing exercises (plantar fascia, plantar flexor muscles)
  Arms: Physiotherapy group
Other: Mobilization — Antero-posterior gliding, talocrural traction, metatarsal mobilization
  Arms: Home exercise group; Physiotherapy group

SUMMARY:
Plantar fasciitis is seen common in clinics and responsible from most of foot related pain problems. There are many treatment modalities in the literature as well as there is no golden standard to treat plantar fasciitis in non-surgical ways. The aim of this study is to compare intensive physiotherapy program, home based exercise program and control group decide the most effective rehabilitation program in plantar fasciitis.

DETAILED DESCRIPTION:
Plantar fasciitis is frequently seen in adult population as a pain related problem of the foot. Pain, as a most prominent symptom, is caused from repetitive microtraumas and inflammation where plantar fascia attaches to the calcaneus. Pain starts from heel pad or medial tubercule of the calcaneus and spreads through plantar fascia and medial longitudinal arch.

Obesity, increased foot pronation, difference in extremity length, long standing duration and Achilles tendon tightness are some of the factors which stress plantar fascia and sometimes cause degenerative changes on it. Weakness of intrinsic muscle is also another factor which is thought to be related with plantar fasciitis.

Diagnosis is mostly depends on history and physical examination. First steps in the morning, walking after long rest, and palpation of medial tubercule of calcaneus are painful.

According to the literature, non-surgical treatment modalities relieve symptoms of patients successfully. Orthotics, night splints, manipulation interventions with conventional methods are effective to decrease pain and improve function. There are various physiotherapy treatment approaches in plantar fasciitis but there is no consensus about most effective treatment program. Stretching of plantar flexor muscles and plantar fascia is one of the core elements of the treatment plan. Strengthening exercises together with stretching were shown more effective than only stretching. Foot orthoses are thought to prevent increased pronation and relieving stress on plantar fascia in patients with plantar fasciitis. Usage of insoles with night splints is found more effective. Taping is also helpful to acute pain control. Short foot exercises as isolated intrinsic foot muscles strengthening helps to providing subtalar foot position and supports plantar fascia and foot arches. Manual techniques improve lower extremity joint mobility and decreases related pain. Extracorporeal Shock Wave Therapy is suggested to try after at least six month ineffective conservative treatments. If symptoms resist more than six months and non-conservative treatments are found ineffective, invasive approaches as steroid injections are applicable.

Treatment of this common problem in population is important to ensure patients returning in earliest period to daily life with full physical capacity. There are many conservative options to treat plantar fasciitis but best treatment program combination was not clear The aim of this study is to compare intensive physiotherapy program, home based exercise program and control group decide the most effective rehabilitation program in plantar fasciitis.

ELIGIBILITY:
Inclusion Criteria:

Older than 18 years, Baseline Roles and Maudsley score > 2, Accepting and signing consent form Daily usage of insoles which was prescribed by doctor No history of systemic disease and surgery that affects foot biomechanics No history of cognitive, mental, neurological or psychological problems.

Exclusion Criteria:

Presence of chronic or active infection in treatment site, Not accepting to participate in the study Systemic, neurologic, rheumatologic,and vascular disease history, Pregnancy, BMI > 35 kg/m2, History of foot and/or ankle surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2018-07-15 (Actual); Primary Completion 2019-12-15 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
Perception of pain | 6 weeks
  Perception of pain with Visual Analog Scale (VAS) with palpation, first steps in the morning and after long walk.
  The Visual Analog Scale is a valid and reliable measure of pain intensity. To rate pain intensity a mark is placed on a 100-mm VAS. The VAS is horizontally positioned with the extremes labeled''least possible pain'' and ''worst possible pain. Using a ruler, the score is determined by measuring the distance (mm) on the 100 mm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Subjects will be asked to rate pain in three different conditions as palpation, first steps in the morning and after long walk.

SECONDARY OUTCOMES:
Perception of quality of life | 6 weeks
  The World Health Organization (WHO) Quality of Life - Bref Questionnaire is a 26-item self-administered instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items. Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100-scale. Higher score presents better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Nilgun BEK, PT, PhD, Professor, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pfeffer G, Bacchetti P, Deland J, Lewis A, Anderson R, Davis W, Alvarez R, Brodsky J, Cooper P, Frey C, Herrick R, Myerson M, Sammarco J, Janecki C, Ross S, Bowman M, Smith R. Comparison of custom and prefabricated orthoses in the initial treatment of proximal plantar fasciitis. Foot Ankle Int. 1999 Apr;20(4):214-21. doi: 10.1177/107110079902000402. PMID 10229276
- [Background] Goff JD, Crawford R. Diagnosis and treatment of plantar fasciitis. Am Fam Physician. 2011 Sep 15;84(6):676-82. PMID 21916393
- [Background] Podolsky R, Kalichman L. Taping for plantar fasciitis. J Back Musculoskelet Rehabil. 2015;28(1):1-6. doi: 10.3233/BMR-140485. PMID 24867905
- [Background] Thomas JL, Christensen JC, Kravitz SR, Mendicino RW, Schuberth JM, Vanore JV, Weil LS Sr, Zlotoff HJ, Bouche R, Baker J; American College of Foot and Ankle Surgeons heel pain committee. The diagnosis and treatment of heel pain: a clinical practice guideline-revision 2010. J Foot Ankle Surg. 2010 May-Jun;49(3 Suppl):S1-19. doi: 10.1053/j.jfas.2010.01.001. PMID 20439021
- [Background] Martin RL, Davenport TE, Reischl SF, McPoil TG, Matheson JW, Wukich DK, McDonough CM; American Physical Therapy Association. Heel pain-plantar fasciitis: revision 2014. J Orthop Sports Phys Ther. 2014 Nov;44(11):A1-33. doi: 10.2519/jospt.2014.0303. PMID 25361863
- [Background] Digiovanni BF, Nawoczenski DA, Malay DP, Graci PA, Williams TT, Wilding GE, Baumhauer JF. Plantar fascia-specific stretching exercise improves outcomes in patients with chronic plantar fasciitis. A prospective clinical trial with two-year follow-up. J Bone Joint Surg Am. 2006 Aug;88(8):1775-81. doi: 10.2106/JBJS.E.01281. PMID 16882901
- [Background] Sweeting D, Parish B, Hooper L, Chester R. The effectiveness of manual stretching in the treatment of plantar heel pain: a systematic review. J Foot Ankle Res. 2011 Jun 25;4:19. doi: 10.1186/1757-1146-4-19. PMID 21703003
- [Background] Cheung RT, Sze LK, Mok NW, Ng GY. Intrinsic foot muscle volume in experienced runners with and without chronic plantar fasciitis. J Sci Med Sport. 2016 Sep;19(9):713-5. doi: 10.1016/j.jsams.2015.11.004. Epub 2015 Nov 22. PMID 26655866
- [Background] Moon DC, Kim K, Lee SK. Immediate Effect of Short-foot Exercise on Dynamic Balance of Subjects with Excessively Pronated Feet. J Phys Ther Sci. 2014 Jan;26(1):117-9. doi: 10.1589/jpts.26.117. Epub 2014 Feb 6. PMID 24567688
- [Background] McKeon PO, Fourchet F. Freeing the foot: integrating the foot core system into rehabilitation for lower extremity injuries. Clin Sports Med. 2015 Apr;34(2):347-61. doi: 10.1016/j.csm.2014.12.002. Epub 2015 Jan 24. PMID 25818718
- [Background] Bennett PJ, Patterson C, Wearing S, Baglioni T. Development and validation of a questionnaire designed to measure foot-health status. J Am Podiatr Med Assoc. 1998 Sep;88(9):419-28. doi: 10.7547/87507315-88-9-419. PMID 9770933